CLINICAL TRIAL: NCT00075582
Title: Vincristine, Dactinomycin, and Lower Doses of Cyclophosphamide With or Without Radiation Therapy for Patients With Newly Diagnosed Low-Risk Embryonal/Botryoid/Spindle Cell Rhabdomyosarcoma
Brief Title: Vincristine, Dactinomycin, and Cyclophosphamide With or Without Radiation Therapy in Treating Patients With Newly Diagnosed Low-Risk Rhabdomyosarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARST0331; NCI-2009-00425 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ARST0331 (Other: Children's Oncology Group); CDR0000347078 (Other: Clinical Trials.gov); U10CA098543 (NIH)
Record Dates: First submitted 2004-01-09; First posted 2004-01-12 (Estimated); Results first posted 2014-04-11 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Adult Rhabdomyosarcoma; Embryonal Childhood Rhabdomyosarcoma; Embryonal-botryoid Childhood Rhabdomyosarcoma; Previously Untreated Childhood Rhabdomyosarcoma
MeSH Terms: conditions — Rhabdomyosarcoma | interventions — Surgical Procedures, Operative; Congresses as Topic; Dactinomycin; Cyclophosphamide; Vincristine; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regimen I (chemotherapy, radiotherapy) (Experimental): Patients receive VAC chemotherapy comprising vincristine sulfate IV over 1 minute on day 1 of weeks 1-9 and dactinomycin IV over 1 minute and cyclophosphamide IV over 1 hour on day 1 of weeks 1, 4, 7, and 10; VA chemotherapy comprising vincristine sulfate IV over 1 minute on day 1 of weeks 13-21 and dactinomycin IV over 1 minute on day 1 of weeks 13, 16, 19, and 22 (dactinomycin is omitted during radiation therapy); and radiation therapy, 5 days a week, beginning on week 13 and continuing for 4-7 weeks, depending on prescribed dose. Some patients do not receive radiation therapy; some start it at week 24. (closed to accrual as of 08/13/2010)
  Interventions: Drug: dactinomycin; Drug: cyclophosphamide; Drug: vincristine sulfate; Radiation: radiation therapy
- Regimen II (chemotherapy, radiotherapy, surgery) (Experimental): Patients receive VAC chemotherapy and radiation therapy as in regimen I and VA chemotherapy comprising vincristine sulfate IV over 1 minute on day 1 of weeks 13-21, 25-33, and 37-45 and dactinomycin IV over 1 minute on day 1 of weeks 13, 16, 19, 22, 25, 28, 31, 34, 37, 40, 43, and 46 (dactinomycin is omitted during radiation therapy). Some patients do not receive radiation therapy; some start it at week 13 and some at week 24. Some patients have conventional surgery (second-look) at Week 13 (closed to accrual as of 9/23/2011).
  Interventions: Procedure: conventional surgery; Drug: dactinomycin; Drug: cyclophosphamide; Drug: vincristine sulfate; Radiation: radiation therapy

INTERVENTIONS:
Procedure: conventional surgery — Some patients may undergo second-look surgery
  Other Names: surgery, conventional
  Arms: Regimen II (chemotherapy, radiotherapy, surgery)
Drug: dactinomycin — Given IV
  Other Names: ACT-D; actinomycin C1; AD; Cosmegen; DACT
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: vincristine sulfate — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
Radiation: radiation therapy — Undergo radiotherapy
  Other Names: irradiation; radiotherapy; therapy, radiation

SUMMARY:
This phase III trial is studying how well combination chemotherapy and radiation therapy work in treating patients with newly diagnosed low-risk rhabdomyosarcoma. Drugs used in chemotherapy, such as vincristine, dactinomycin, and cyclophosphamide, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy may kill more tumor cells. It is not yet known which treatment regimen is more effective in treating low-risk rhabdomyosarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the failure-free survival of patients with newly diagnosed low-risk rhabdomyosarcoma treated with vincristine (V), dactinomycin (A), cyclophosphamide (C), and radiotherapy.

SECONDARY OBJECTIVES:

I. Determine local control rates in patients treated with this regimen. II. Determine the rate of second-look surgery in patients with bulk residual tumor at diagnosis (clinical group III) and the proportion of second-look surgeries that render patients treated with this regimen tumor-free or with microscopic tumor only and evaluate the pathologic significance of that residual tumor.

III. Determine the local control rates in patients with clinical group III disease treated with response-adjusted radiotherapy doses after second-look surgical resection.

OUTLINE: This is a nonrandomized, multicenter study. Patients are assigned to 1 of 2 treatment regimens according to disease stage and clinical group.

REGIMEN I (subset 1 patients) [closed to accrual as of 08/13/2010: Patients receive VAC chemotherapy comprising vincristine IV over 1 minute on day 1 of weeks 1-9 and dactinomycin IV over 1 minute and cyclophosphamide IV over 1 hour on day 1 of weeks 1, 4, 7, and 10; VA chemotherapy comprising vincristine IV over 1 minute on day 1 of weeks 13-21 and dactinomycin* IV over 1 minute on day 1 of weeks 13, 16, 19, and 22; and radiotherapy**, 5 days a week, beginning on week 13 and continuing for 4-7 weeks, depending on prescribed dose.

REGIMEN II (subset 2 patients)[closed to accrual as of 9/23/2011]: Patients receive VAC chemotherapy and radiotherapy** as in regimen I and VA chemotherapy comprising vincristine IV over 1 minute on day 1 of weeks 13-21, 25-33, and 37-45 and dactinomycin* IV over 1 minute on day 1 of weeks 13, 16, 19, 22, 25, 28, 31, 34, 37, 40, 43, and 46. Patients with clinical group III disease may undergo second-look surgery at week 13 followed by response-adjusted radiotherapy, and continued VA* chemotherapy. In both regimens, treatment continues in the absence of disease progression or unacceptable toxicity.

NOTE: *For both regimens, dactinomycin is omitted during radiotherapy.

NOTE: **Clinical Group I tumors and those with Clinical Group III uterine/cervix primary disease with negative nodes who have undergone a complete resection (i.e. hysterectomy) at Week 13 do not receive radiotherapy at Week 13

Patients are followed up every 3 months for 1 year, every 4 months for 2 years, every 6 months for 1 year, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed newly diagnosed embryonal rhabdomyosarcoma (RMS), botryoid or spindle cell variants of embryonal RMS, or embryonal ectomesenchymoma, meeting criteria for 1 of the following subsets:

  * Subset 1, defined by meeting 1 of the following criteria (closed to accrual as of 08/13/2010):

    * Stage 1 and clinical group I (completely resected) or II (microscopic residual disease and/or regional lymph node involvement) disease
    * Stage 1 and clinical group III (gross residual disease) disease arising in the orbit
    * Stage 2 and clinical group I or II disease
  * Subset 2, defined by meeting 1 of the following criteria (closed to accrual as of 09/23/2011):

    * Stage 1 and clinical group III disease arising in a non-orbit site
    * Stage 3 and clinical group I or II disease
* Prior staging ipsilateral retroperitoneal lymph node dissection required for all patients age 10 and over with paratesticular tumors and patients under 10 years of age with clinically or radiographically involved lymph nodes (except when extensive lymph node involvement is identified by imaging studies)

  * If there is extensive gross node involvement only confirmatory node biopsy is recommended and the patient is classified as Clinical Group III
* Prior regional lymph node sampling required for patients with extremity tumors
* None of the following diagnoses:

  * Intermediate-risk embryonal RMS
  * Metastatic embryonal RMS
  * Alveolar RMS
  * Undifferentiated sarcoma
  * RMS not otherwise specified (NOS)
  * Other soft tissue sarcoma, including sarcoma NOS
* Prior enrollment on clinical trial COG-D9902
* Performance status - ECOG 0-2
* Performance status - Karnofsky 50-100% (≥ 16 years old)
* Performance status - Lansky 50-100% (< 16 years old)
* Absolute neutrophil count at least 750/mm^3
* Platelet count at least 75,000/mm^3 (transfusion independent)
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)*
* Creatinine* based on age/gender as follows:

  * No greater than 0.8 mg/dL for patients age 5 and under
  * No greater than 1.0 mg/dL for patients age 6 to 9
  * No greater than 1.2 mg/dL for patients age 10 to 12
  * No greater than 1.4 mg/dL for female patients age 13 and over
  * No greater than 1.5 mg/dL for male patients age 13 to 15
  * No greater than 1.7 mg/dL for male patients age 16 and over
* Creatinine clearance* or radioisotope glomerular filtration rate at least 70 mL/min/1.73 m^2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infection
* No prior chemotherapy (except for patients treated on the related intermediate-risk study)
* Prior steroids allowed
* No prior radiotherapy

Max Age: 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 390 (Actual)
Dates: Start 2004-09-04; Primary Completion 2012-08-13 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Walterhouse, MD, Principal Investigator — Children's Oncology Group
Locations (163):
- United States (138):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Children's Oncology Group, Arcadia, California
  - Southern California Permanente Medical Group, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Childrens Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - University of California San Francisco Medical Center-Parnassus, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Memorial Healthcare System - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic - Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - M D Anderson Cancer Center- Orlando, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph Children's Hospital of Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - University of Illinois, Chicago, Illinois
  - Childrens Memorial Hospital, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Raymond Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital-Main Campus, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Michigan State University - Breslin Cancer Center, Lansing, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - UMDNJ - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospitals Inc, Asheville, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Presbyterian Hospital, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Medical Center of Dayton, Dayton, Ohio
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Childrens Hospital-King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - West Virginia University Charleston, Charleston, West Virginia
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (7):
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Sydney, New South Wales
  - Sydney West Area Health Service-Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (13):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - Chedoke-McMaster Hospitals, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Hospital Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Ste-Foy, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- San Jorge Children's Hospital, Santurce, Puerto Rico
- Switzerland (2):
  - Swiss Pediatric Oncology Group - Geneva, Geneva
  - Swiss Pediatric Oncology Group - Lausanne, Lausanne

REFERENCES:
- [Background] Woolson RF (1981) Rank-tests and a one-sample log-rank test for comparing observed survival-data to a standard population. Biometrics 37: 687-696.
- [Derived] Proia AD. Spindle Cell/Sclerosing Rhabdomyosarcoma of the Orbit. Ophthalmic Plast Reconstr Surg. 2023 Jan-Feb 01;39(1):e17-e20. doi: 10.1097/IOP.0000000000002252. Epub 2022 Jul 13. PMID 35829629
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Regimen I (Chemotherapy, Radiotherapy) | Regimen II (Chemotherapy, Radiotherapy, Surgery)
Started | 305 | 85
Completed | 255 | 50
Not Completed | 50 | 35
Not completed — Adverse Event | 3 | 1
Not completed — Lack of Efficacy | 4 | 8
Not completed — Physician Decision | 5 | 8
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Ineligible for study | 36 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen I (Chemotherapy, Radiotherapy) | Regimen II (Chemotherapy, Radiotherapy, Surgery) | Total
Number analyzed (Participants) | 305 | 85 | 390
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.69 (5.81) | 5.02 (6.78) | 7.11 (6.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 55 | 143
  Male | 217 | 30 | 247
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 9 | 2 | 11
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 39 | 9 | 48
  White | 228 | 65 | 293
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 26 | 7 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 9 | 47
  Not Hispanic or Latino | 255 | 71 | 326
  Unknown or Not Reported | 12 | 5 | 17
Region of Enrollment [Number; unit: participants]
  United States | 269 | 77 | 346
  Canada | 21 | 5 | 26
  Australia | 7 | 3 | 10
  Netherlands | 2 | 0 | 2
  New Zealand | 1 | 0 | 1
  Puerto Rico | 2 | 0 | 2
  Switzerland | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Low-risk Rhabdomyosarcoma in Subset 1 Failure Free at 5 Years Following Study Entry
Description: Kaplan Meier estimate of failure free survival at 5 years, where failure free survival is defined as the time to relapse, progression, second malignancy, and death whichever occurs first.
Time Frame: From enrollment up to 5 years
Population: Patients found not to meet the eligibility requirements are by group policy not followed for adverse events or outcome.
Measure: Number (95% Confidence Interval); unit: Estimated percentage of participants
Arm/Group | Regimen I (Chemotherapy, Radiotherapy) | Regimen II (Chemotherapy, Radiotherapy, Surgery)
Number analyzed (Participants) | 269 | 69
Estimated percentage of participants | 87 [82 to 91] | 67 [52 to 79]

2. Primary Outcome: Percentage of Patients With Stage 1, Clinical Group IIB or C (Node Positive) or Stage 2 Failure Free at 5 Years Following Study Entry
Description: as for outcome 1
Time Frame: From enrollment up to 5 years
Population: All eligible patients among this subset of regimen 1 patients were included in this outcome measure restricted to regimen 1 patients (there were 36 patients determined ineligible). Patients found not to meet the eligibility requirements are by group policy not followed for adverse events or outcome measures.
Measure: Number (95% Confidence Interval); unit: Estimated percentage of participants
Arm/Group | Regimen I (Chemotherapy, Radiotherapy)
Number analyzed (Participants) | 30
Estimated percentage of participants | 90 [72 to 97]

3. Primary Outcome: Percentage of Patients With Low-risk Rhabdomyosarcoma in Subset 2 Failure Free at 5 Years Following Study Entry
Description: as for outcome 1
Time Frame: From enrollment up to 5 years
Population: All eligible patients among this subset of regimen 2 patients were included in this outcome measure to regimen 2 patients (there were 16 patients determined ineligible). Patients found not to meet the eligibility requirements are by group policy not followed for adverse events or outcome measures.
Measure: Number (95% Confidence Interval); unit: Estimated percentage of participants
Arm/Group | Regimen II (Chemotherapy, Radiotherapy, Surgery)
Number analyzed (Participants) | 69
Estimated percentage of participants | 67 [52 to 79]

4. Secondary Outcome: Cumulative Incidence of Patients Who Receive Reduced Doses of Radiation Therapy
Description: The local failure rate will be estimated using cumulative incidence curves.
Time Frame: From enrollment up to 5 years
Population: Patients who received reduced doses of radiation therapy.
Measure: Number (95% Confidence Interval); unit: stimated percentage of participants
Groups:
- Regimen I (Chemotherapy, Radiotherapy): Stage I/II group IIA patients receive VAC chemotherapy comprising vincristine sulfate IV over 1 minute on day 1 of weeks 1-9 and dactinomycin IV over 1 minute and cyclophosphamide IV over 1 hour on day 1 of weeks 1, 4, 7, and 10; VA chemotherapy comprising vincristine sulfate IV over 1 minute on day 1 of weeks 13-21 and dactinomycin IV over 1 minute on day 1 of weeks 13, 16, 19, and 22 (dactinomycin is omitted during radiation therapy); and radiation therapy, 5 days a week, beginning on week 13 and continuing for 4-7 weeks, depending on prescribed dose. Some patients do not receive radiation therapy; some start it at week 24. (closed to accrual as of 08/13/2010)
  dactinomycin: Given IV
  cyclophosphamide: Given IV
  vincristine sulfate: Given IV
  radiation therapy: Undergo radiotherapy
- Regimen II (Chemotherapy, Radiotherapy, Surgery): Group III patients with orbit primary receive VAC chemotherapy comprising vincristine sulfate IV over 1 minute on day 1 of weeks 1-9 and dactinomycin IV over 1 minute and cyclophosphamide IV over 1 hour on day 1 of weeks 1, 4, 7, and 10; VA chemotherapy comprising vincristine sulfate IV over 1 minute on day 1 of weeks 13-21 and dactinomycin IV over 1 minute on day 1 of weeks 13, 16, 19, and 22 (dactinomycin is omitted during radiation therapy); and radiation therapy, 5 days a week, beginning on week 13 and continuing for 4-7 weeks, depending on prescribed dose. Some patients do not receive radiation therapy; some start it at week 24. (closed to accrual as of 08/13/2010)
  dactinomycin: Given IV
  cyclophosphamide: Given IV
  vincristine sulfate: Given IV
  radiation therapy: Undergo radiotherapy
Arm/Group | Regimen I (Chemotherapy, Radiotherapy) | Regimen II (Chemotherapy, Radiotherapy, Surgery)
Number analyzed (Participants) | 52 | 62
stimated percentage of participants | 0.081 [0.046 to 0.116] | 0.115 [0.035 to 0.195]

5. Secondary Outcome: Percentage of Patients With Delayed Surgical Procedures
Description: The decision to perform second-look surgery should be based on the physical examination and imaging studies at Week 12 and should only be considered if a reasonable functional and cosmetic result is anticipated.
Time Frame: At 13 weeks after induction
Population: All eligible Stage I Group III nonorbit primary and stage III group I/II patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Regimen II (Stage I Group III Nonorbit or Stage III Group I/II: Stage I group III nonorbit primary or stage III group I/II patients receive VAC chemotherapy comprising vincristine sulfate IV over 1 minute on day 1 of weeks 1-9 and dactinomycin IV over 1 minute and cyclophosphamide IV over 1 hour on day 1 of weeks 1, 4, 7, and 10; VA chemotherapy comprising vincristine sulfate IV over 1 minute on day 1 of weeks 13-21 and dactinomycin IV over 1 minute on day 1 of weeks 13, 16, 19, and 22 (dactinomycin is omitted during radiation therapy); and radiation therapy, 5 days a week, beginning on week 13 and continuing for 4-7 weeks, depending on prescribed dose. Some patients do not receive radiation therapy; some start it at week 24. (closed to accrual as of 08/13/2010)
  dactinomycin: Given IV
  cyclophosphamide: Given IV
  vincristine sulfate: Given IV
  radiation therapy: Undergo radiotherapy
Arm/Group | Regimen II (Stage I Group III Nonorbit or Stage III Group I/II
Number analyzed (Participants) | 45
percentage of participants | 0.49 [0.34 to 0.64]

6. Secondary Outcome: Cumulative Incidence of Group III Patients Who Received With Reduced Radiotherapy Dose
Description: The local failure rate will be estimated using cumulative incidence curves for Group III patients who received reduced doses of radiation therapy after second look surgical resection.
Time Frame: From enrollment up to 20 weeks
Population: Patients with Group III vaginal primary tumor
Measure: Number; unit: Estimated percentage of participants
Arm/Group | Regimen II (Stage I Group III Nonorbit or Stage III Group I/II
Number analyzed (Participants) | 5
Estimated percentage of participants | 0

ADVERSE EVENTS:
Description: Patients found not to meet the eligibility requirements are by group policy not followed for adverse events or outcome.
Arm/Group | Regimen I (Chemotherapy, Radiotherapy) | Regimen II (Chemotherapy, Radiotherapy, Surgery)
Serious Adverse Events (participants affected / at risk) | 1/272 | 1/70
Other Adverse Events (participants affected / at risk) | 74/272 | 27/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen I (Chemotherapy, Radiotherapy) (N=272) | Regimen II (Chemotherapy, Radiotherapy, Surgery) (N=70)
Neutrophil count decreased (Investigations) | 0 | 1 (1)
White blood cell decreased (Investigations) | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen I (Chemotherapy, Radiotherapy) (N=272) | Regimen II (Chemotherapy, Radiotherapy, Surgery) (N=70)
Anemia (Blood and lymphatic system disorders) | 14 (14) | 9 (9)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 14 (14) | 7 (7)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0
Photophobia (Eye disorders) | 1 (1) | 0
Watering eyes (Eye disorders) | 1 (1) | 0
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0
Flatulence (Gastrointestinal disorders) | 1 (1) | 0
Ileus (Gastrointestinal disorders) | 1 (1) | 0
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 0
Oral pain (Gastrointestinal disorders) | 1 (1) | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 0
Facial pain (General disorders) | 1 (1) | 0
Fatigue (General disorders) | 1 (1) | 0
Fever (General disorders) | 5 (5) | 4 (4)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 1 (1)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 2 (2) | 0 (0)
Catheter related infection (Infections and infestations) | 2 (2) | 1 (1)
Conjunctivitis infective (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 4 (4) | 5 (5)
Rhinitis infective (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 9 (9) | 2 (2)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 7 (7) | 3 (3)
Blood bilirubin increased (Investigations) | 2 (2) | 0
Creatinine increased (Investigations) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2) | 3 (3)
Neutrophil count decreased (Investigations) | 43 (43) | 15 (15)
Platelet count decreased (Investigations) | 10 (10) | 1 (1)
Weight loss (Investigations) | 2 (2) | 3 (3)
White blood cell decreased (Investigations) | 23 (23) | 10 (10)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Headache (Nervous system disorders) | 1 (1) | 0
Peripheral motor neuropathy (Nervous system disorders) | 4 (4) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4) | 1 (1)
Pyramidal tract syndrome (Nervous system disorders) | 1 (1) | 0
Scrotal pain (Reproductive system and breast disorders) | 1 (1) | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (3) | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0
Vascular disorders - Other (Vascular disorders) | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.